CLINICAL TRIAL: NCT00503087
Title: Evaluation of Pain Reduction in the Administration of Saline Injections by the Usage of Pneumatic Skin Flattening (PSF)
Brief Title: Evaluation of Pain Reduction in the Administration of Saline Injections by the Usage of Pneumatic Skin Flattening
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PalJect Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TASMC 07- TL -268 CTIL
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: Injections; Vacuum; Pain; Pneumatic Skin Flattening; PSF
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Saline Injection
Device: Pneumatic Skin Flattening (PSF)

SUMMARY:
Each participant will be administered 2 injections of saline - the first in the right gluteal area and the second in the left gluteal area. Both injections will be administered intra-muscularly by the same clinician. One injection will be given with vacuum (Pneumatic Skin Flattening or PSF Machine) and the other without vacuum. The order of the injections will be randomly assigned. Each subject will serve as a control for himself. Between injections a 30 min pause will be given to minimize pain sensation bias of the previous injection. Immediately after each injection the pain level will be assessed by the VAS scale. The researcher assessing the pain will be blinded for the type of injection given. The evaluation of the pain reduction will be made by comparison of the pain level with and without the application of the PSF.

Hypothesis: PSF Technique will reduce the pain associated with saline injections.

DETAILED DESCRIPTION:
Injections are currently the gold-standard for administrating various medications parenterally. The most significant side-effect related to injections is the accompanying pain. Injection pain is related to the penetration of the skin by the needle and to the mechanical and chemical effects of the drug during and after its injection. This pain remains a major obstacle in medication administration in children as well as in other populations subject to needle-phobia because of the pain experience. The associated pain may thus prevent optimized medical care for these patients.

Current methods to alleviate immediate pain include the utilization of topical anesthesia whereas some patients do not utilize any form of pain relief and simply endure the pain of the injection. Other methods for pain reduction are taking advantage of the applying pressure or vibration to alleviate pain. These methods have resulted in a number of pain relieving devices currently on the market. Such predicate devices primarily involve vibration devices commonly used to alleviate the injection pain. Published data suggests possible use of pressure application mechanism in pain alleviation related to injections.

We suggest here, for the first time, the use of the Pneumatic Skin Flattening (PSF) technology for alleviation of pain associated with injections. The PSF technology is currently used worldwide in the FDA cleared Serenity device (Serenity, Inolase Ltd.) for pain reduction in hair removal. The device generates contact and compression between a transparent sapphire window and the skin. The compression creatures pressure signal which, based on the gate theory, is though to depress the pain associated with the hair removal treatment. We assume the same mechanism would apply for the reduction of pain associated with injections.

Comparison: Intra-Subject pain level change of injection with PSF and without PSF

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Healthy
* Patient informed consent must be obtained

Exclusion Criteria:

* Pregnant or nursing women
* Patients unable to understand or sign the informed consent form
* Anticoagulant or aspirin treatment
* Subjects with a history of vaso-vagal reactions to injections
* Coagulopathies
* Skin disease
* Chronic usage of medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-08; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
VAS pain scaling differences between saline injection with PSF and without PSF | Immediately after each injection

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Halpern, MD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Emergency Department- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] MELZACK R, WALL PD. On the nature of cutaneous sensory mechanisms. Brain. 1962 Jun;85:331-56. doi: 10.1093/brain/85.2.331. No abstract available. PMID 14472486
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Lask G, Friedman D, Elman M, Fournier N, Shavit R, Slatkine M. Pneumatic skin flattening (PSF): a novel technology for marked pain reduction in hair removal with high energy density lasers and IPLs. J Cosmet Laser Ther. 2006 Jun;8(2):76-81. doi: 10.1080/14764170600719775. PMID 16766485